CLINICAL TRIAL: NCT02000674
Title: Succinylcholine vs Rocuronium for Prehospital Emergency Intubation : a Randomized Trial
Brief Title: Succinylcholine vs Rocuronium for Prehospital Emergency Intubation
Acronym: CURASMUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Unité de Soutien Méthodologique (CHU de La Réunion) (Unknown); SAMU de Paris, Hôpital Necker - Enfants Malades (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/CHU/05; 2013-001438-16 (EudraCT Number)
Record Dates: First submitted 2013-10-09; First posted 2013-12-04 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-03

CONDITIONS: Coma; Major Trauma; Respiratory Distress; Shock
Keywords: tracheal intubation; pre hospital emergency
MeSH Terms: conditions — Coma; Dyspnea; Shock | interventions — Succinylcholine; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Administration of Succinylcholine (Active Comparator): Intubation after IV administration of Succinylcholine 1mg/kg
  Interventions: Drug: Succinylcholine : 1mg/kg
- Administration of Rocuronium (Experimental): Intubation after IV administration of Rocuronium 1.2 mg/kg
  Interventions: Drug: Rocuronium : 1.2 mg/kg

INTERVENTIONS:
Drug: Succinylcholine : 1mg/kg
  Other Names: Suxaméthonium Aguetant®; SUXAMETHONIUM BIOCODEX 50 mg/ml, solution injectable
  Arms: Administration of Succinylcholine
Drug: Rocuronium : 1.2 mg/kg
  Other Names: ESMERON®
  Arms: Administration of Rocuronium

SUMMARY:
All adult patients with spontaneous cardiac activity and requiring tracheal intubation in the pre hospital emergency context will be included in order to compare the use of succinylcholine vs Rocuronium for prehospital emergency intubation.

DETAILED DESCRIPTION:
All adult patients with spontaneous cardiac activity and requiring tracheal intubation in the pre hospital emergency context will be included. All intubation will be performed by an emergency physician or a nurse specialized in anesthesia. For patients with spontaneous cardiac activity, rapid sequence intubation will be performed to allow intubation.

Comparisons studied will be : Intubation success rate at the first laryngoscopy, glottis exposure assessed by Cormack and Lehane classification, difficult intubation rate assessed by the Intubation Difficult Score (IDS), the conditions of intubation assessed by the Copenhagen score, the need for alternative airway techniques and the immediate post intubation complications rate as vomiting, dental trauma, pulmonary inhalation, arterial desaturation , hypotension episodes and cardiac arrest occurrence.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with spontaneous cardiac activity and requiring tracheal intubation in the pre hospital emergency context

Exclusion Criteria:

* Patients in cardiac arrest;
* Patients under-18s;
* Patients under guardianship ;
* Pregnancy known;
* Patients with cons to one of the following three drugs: rocuronium, succinylcholine, sugammadex;
* Patients not affiliated to a social security scheme (beneficiary or legal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1321 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
First-pass intubation success rate | between 1 hour to 3 hours after inclusion
  Measured by the proportion of successful intubation in the first laryngoscopy.

SECONDARY OUTCOMES:
Incidence of difficult intubation | between 1 hour to 3 hours after inclusion
  measured by the Intubation Difficulty Scale
Intubation conditions assessment | between 1 hour to 3 hours after inclusion
  using the Copenhagen score
Need for alternate airway devices | between 1 hour to 3 hours after inclusion
early intubation-related complications | between 1 hour to 3 hours after inclusion
  complications : esophageal intubation, mainstem intubation, vomiting, pulmonary aspiration, dental trauma, bronchospasm or laryngospasm, ventricular tachycardia, arterial desaturation, hypotension, or cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Combes, MD, Principal Investigator — CHU de La Réunion
Locations (17):
- France (17):
  - CHU de La Réunion, Saint-Denis, La Réunion
  - CHU de la Réunion, Saint-Pierre, La Réunion
  - CHU Avicenne, Bobigny
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU Raymond Poincaré, Garches
  - CH Gonesse, Gonesse
  - CHRU de Lille, Lille
  - CH Marc Jacquet, Melun
  - CHU de Nîmes, Nîmes
  - CHU Hôtel-Dieu, Paris
  - CHU Lariboisière, Paris
  - CHU Necker, Paris
  - CHU Pitié-Salpêtrière, Paris
  - CH René Dubos, Pontoise
  - CH Annecy, Pringy
  - CHU Toulouse - Hôpital PURPAN, Toulouse

REFERENCES:
- [Derived] Guihard B, Chollet-Xemard C, Lakhnati P, Vivien B, Broche C, Savary D, Ricard-Hibon A, Marianne Dit Cassou PJ, Adnet F, Wiel E, Deutsch J, Tissier C, Loeb T, Bounes V, Rousseau E, Jabre P, Huiart L, Ferdynus C, Combes X. Effect of Rocuronium vs Succinylcholine on Endotracheal Intubation Success Rate Among Patients Undergoing Out-of-Hospital Rapid Sequence Intubation: A Randomized Clinical Trial. JAMA. 2019 Dec 17;322(23):2303-2312. doi: 10.1001/jama.2019.18254. PMID 31846014